CLINICAL TRIAL: NCT06886594
Title: The Effect of Breast Self Examination Training Using Breast Examination Simulator on Breast Cancer Knowledge Level and Health Beliefs
Brief Title: The Effect of BSE Training on Breast Cancer Knowledge Level and Health Beliefs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Emine Derya Ister, associate professor.Dr., Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: BSEKSU
Record Dates: First submitted 2025-02-19; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Health Behavior; Healthy Female; Education
Keywords: Breast Canser; Self-Breast Examination; Breast cancer knowledge level; health belief
MeSH Terms: conditions — Health Behavior; Breast Self-Examination

STUDY DESIGN:
Intervention Model Description: The content of the training given to the experimental group was prepared in accordance with the "Breast Cancer Prevention, Screening, Diagnosis, Treatment and Follow-up Clinical Guide 2020 (Version 1.0)" of the Ministry of Health of the Republic of Turkey. After the completion of the theoretical training, each woman in the experimental group was given BSE practical training using the demonstration method by the first researcher in line with the steps in the "Breast Self-Examination" brochure prepared by the "Cancer Early Diagnosis, Screening and Training Center of the Ministry of Health of the Republic of Turkey" using the "Wearable Breast Examination Simulator". Then, each woman was provided with the simulator to wear and perform BSE on the model. The application was completed when each woman was provided with BSE correctly. The success indicator of the practical training is that the woman performed the BSE steps correctly as shown in the brochure and detected at least three tumors in
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: triple blinding was done: riple (Participant, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (No Intervention): Procedures Applied to the Control Group
  1. The "Personal Information Form, CHAMPION Health Belief Model Scale, Comprehensive Breast Cancer Knowledge Test" was applied to the control group as a pre-test and three months later as a post-test.
  2. The "Breast Self-Examination" was given to the control group after completing the study.
- Experimental group (Other): 1. Pre-test data were collected by the interviewer using the "Personal Information Form, CHAMPION Health Belief Model Scale, Comprehensive Breast Cancer Knowledge Test" before the training for the experimental group. 2. The breast cancer education program for the experimental group was conducted by the first researcher, and the researcher completed her doctorate in Obstetrics, Women's Health and Diseases Nursing. The content of the education given to the experimental group was prepared in accordance with the Ministry of Health of the Republic of Turkey "Breast Cancer Prevention, Screening, Diagnosis, Treatment and Follow-up Clinical Guide 2020 (Version 1.0)". Each woman in the experimental group was given face-to-face individual education in line with the prepared training material by the first researcher, and their questions were answered at the end of the training.
  Interventions: Other: breast cancer education program training

INTERVENTIONS:
Other: breast cancer education program training — The first researcher conducted the breast cancer education program for the experimental group, and the researcher completed her doctorate in Obstetrics, Gynecology and Diseases Nursing. The content of the education given to the experimental group was prepared in accordance with the "Breast Cancer Prevention, Screening, Diagnosis, Treatment and Follow-up Clinical Guide 2020 (Version 1.0)" of the Ministry of Health of the Republic of Turkey. Each woman in the experimental group was given face-to-face individual education in accordance with the education material prepared by the first researcher, and their questions were answered at the end of the education. After the theoretical education was completed, each woman in the experimental group was given BSE practical education using the "Wearable Breast Examination Simulator" by the first researcher using the demonstration method in accordance with the steps in the "Breast Self-Examination" brochure by the "Cancer Early Diagnosis, Screening
  Arms: Experimental group

SUMMARY:
This study was conducted to evaluate the effects of breast cancer and BSE education given to women aged 40 and over using a breast examination simulator on women's breast cancer knowledge levels and health beliefs. Data were collected in the study using the "Personal Information Form, CHAMPION Health Belief Model Scale, Comprehensive Breast Cancer Knowledge Test". A breast cancer education program was applied to the women in the experimental group. The content of the education given to the experimental group was prepared in accordance with the "Breast Cancer Prevention, Screening, Diagnosis, Treatment and Follow-up Clinical Guide 2020 (Version 1.0)" of the Ministry of Health of the Republic of Turkey. After the completion of the theoretical education, each woman in the experimental group was given BSE practical training using the "Wearable Breast Examination Simulator" by the first researcher in accordance with the steps in the "Breast Self-Examination" brochure by the "Cancer Early Diagnosis, Screening and Education Center of the Ministry of Health of the Republic of Turkey". Then, each woman was provided with the simulator to wear and perform BSE on a model. The application was completed when each woman was able to perform BSE correctly. The success indicator of the practical training was that the woman performed the BSE steps correctly as shown in the brochure and detected at least three tumors in the simulator. The second and third researchers performed the application on the model until each woman in the experimental group performed the procedure steps completely and correctly. The brochure was given to each woman in the experimental group both in print and electronically. A standard reminder message was sent to the experimental group in the 1st, 2nd and 3rd months to perform BSE. Pre-test and post-test data were collected from the control group. No individual in the experimental or control groups was harmed in this study.

DETAILED DESCRIPTION:
Methods Objective This study was conducted to evaluate the effect of the training given to women aged 40 and over on breast cancer and BSE using a breast examination simulator on women's breast cancer knowledge levels and health beliefs.

Type of Study This study is a randomised controlled experimental type. The research was conducted with triple blinding method.

The research data were collected by a trained interviewer independent of the researchers. The women in the experimental and control groups were not informed which group they were included in. The data were analysed by a statistician independent of the researchers.

Research Population-Sample The population of the study consisted of patients aged 40 and over who applied to the gynaecology and obstetrics outpatient clinic of XXX Health Practice and Research Hospital and who met the inclusion criteria of the study. In determining the sample size, the mean and standard deviation values (experiment: 23.97±2.40; control: 25.72±3.51) of the post-test score using Champion's Health Belief Model Scale (CHBMS), which was previously conducted in our country, were used, and the effect size (d) was calculated as 0.58.26 Based on the t test in independent groups, the sample size was calculated as 96 at 95% confidence interval and 80% power criteria. Considering that there may be losses from the study, it was decided to include 100 women in the study.

Inclusion criteria

* Female gender
* Age 40 and over
* At least primary school graduation
* Being open to communication
* Volunteering to participate in the study Exclusion criteria
* Diagnosis of breast cancer
* Receiving training on breast cancer or breast self-examination from health personnel before
* Regular BSE application
* Being a health personnel
* Graduation in the field of health Data Collection Data in the study was collected using the "Personal Information Form, CHAMPION Health Belief Model Scale (CHBMS), Comprehensive Breast Cancer Knowledge Test (BCKT)".

Personal Information Form It consists of questions regarding the sociodemographic characteristics of women and family history of breast cancer. Personal Information Form consists of a total of 10 questions including age, marital status, education level, family history of breast cancer, number of births, breastfeeding status, duration of breastfeeding, and knowledge and practice of breast examination.

Comprehensive Breast Cancer Knowledge Test (BCKT) Comprehensive Breast Cancer Knowledge Test was developed by Stager (1993) in 1993.27 The validity and reliability study of the scale in Turkish was conducted by Başak (2015)28. There are a total of 20 information questions in the scale. The scale is answered as True-False. There are 8 correct and 12 incorrect statements in the questions. There are two dimensions in BCKT: general information and treatability. Questions 1-12 include general information about breast cancer, questions 13-20 include information about the treatability of breast cancer. The Cronbach alpha coefficient of the scale is 0.71.28 In this study, the Cronbach alpha coefficient of BCKT is 0.78.

Champion Health Belief Model Scale (CHBMS) The Health Belief Model, developed by Champion in 1984, consists of six dimensions and 43 items covering six concepts.

Wearable Breast Examination Simulator The Wearable Breast Model (Product code: L50) was used during BSE training so that women could wear it from the front and try to detect masses in the breast model as if it were their own tissue. The model has the features of a visible left nipple depression anomaly and a cellulite image in the left breast tissue, 2 benign tumors that can be felt with palpation examination, 4 malignant tumors, and anomalies that can be felt with palpation examination in the left armpit. This model was used because it was thought that performing breast examination on the woman's own breast would violate the woman's privacy and would not last long. It was also thought that repeated palpation applications as if it were her own breast during the training would increase the courage of women to perform regular BSE.

Research Process Procedures Procedures and Surveys Conducted to the Experimental Group

1. Pre-test data were collected by the interviewer using the "Personal Information Form, CHBMS and BCKT" before the training for the experimental group.
2. The training program for breast cancer was conducted by the first researcher for the experimental group, and the researcher completed her doctorate in Obstetrics, Women's Health and Diseases Nursing. The content of the training given to the experimental group was prepared in accordance with the "Breast Cancer Prevention, Screening, Diagnosis, Treatment and Follow-up Clinical Guide 2020 (Version 1.0)" of the Ministry of Health of the Republic of Turkey.31 Face-to-face individual training was provided to each woman in the experimental group by the first researcher in line with the training material prepared, and their questions were answered at the end of the training.
3. After the completion of the theoretical training, each woman in the experimental group was given BSE practical training using the demonstration method by the first researcher using the "Wearable Breast Examination Simulator" and the steps in the "Breast Self-Examination" brochure of the "Cancer Early Diagnosis, Screening and Training Center of the Ministry of Health of the Republic of Turkey". Then, the second and third researchers had each woman wear the simulator and perform her BSE on the model. The application was completed when each woman performed the BSE correctly. The success indicator of the practical training was that the woman performed the BSE steps correctly as shown in the brochure and detected at least three tumors in the simulator. The second and third researchers had each woman in the experimental group perform the procedure on the model until she performed the procedure steps completely and correctly. The brochure was given to each woman in the experimental group both in print and electronically.
4. A standard reminder message was sent to the experimental group in the 1st, 2nd and 3rd months to perform the BSE. Any questions the women had were answered.
5. Three months after the completion of the Breast Cancer and BSE training program, "CHBMS and BCKT" were applied and the post-test data were collected by the interviewer.

Procedures Performed on the Control Group

1. "Personal Information Form, CHBMS and BCKT" were applied to the control group as a pre-test and three months later as a post-test.
2. The control group was sent a "Breast Self-Examination" informative video and brochure after completing the study

ELIGIBILITY:
Inclusion Criteria:

* Female gender
* Being 40 years old and above
* Being at least a primary school graduate
* Being open to communication
* Being willing to participate in the study

Exclusion Criteria:

* Having a breast cancer diagnosis

  * Having received training from a health care professional on breast cancer or breast self-examination
  * Regular BSE practice
  * Being a health care professional
  * Having a graduation in the health field

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — in terms of breast cancer
Enrollment: 95 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-10-20 (Actual); Study Completion 2025-03-06 (Actual)

PRIMARY OUTCOMES:
Comprehensive Breast Cancer Knowledge Test average score | Baseline-T1
  Scores of women in the experimental and control groups on the Comprehensive Breast Cancer Knowledge Test
Champion Health Belief Model Scale | Baseline-T1
  Champion Health Belief Model Scale mean scores of women in the experimental and control groups
Comprehensive Breast Cancer Knowledge Test average score | 3 months after Baseline-T1
  Scores of women in the experimental and control groups on the Comprehensive Breast Cancer Knowledge Test
Champion Health Belief Model Scale | 3 months after Baseline-T1
  Champion Health Belief Model Scale mean scores of women in the experimental and control groups

CONTACTS AND LOCATIONS:
Locations (1):
- Kahramanmaraş Sütçü İmam Üniversitesi, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Study Protocol — https://bap.ksu.edu.tr/